CLINICAL TRIAL: NCT01278394
Title: An Open-Label, Rising Multiple-Dose, Multi-Center Study to Evaluate the Safety and Efficacy of Topically Applied AN2690 5.0% and 7.5% Solution for the Treatment of Adult Subjects With Onychomycosis of the Great Toenail
Brief Title: Safety and Efficacy Study of Subjects With Onychomycosis of the Great Toenail
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AN2690-ONYC-201; AN2690-ONYC-201 Cohort 3 (Other: Anacor); C3371009 (Other: Pfizer)
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Onychomycosis
Keywords: Onychomycosis; Fungal Nail
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group 1 (Experimental): AN2690 Solution, 5.0%
  Interventions: Drug: AN2690 Solution, 5.0%

INTERVENTIONS:
Drug: AN2690 Solution, 5.0% — Once daily application for 360 days

SUMMARY:
The purpose of the study is to determine the safety and efficacy of 5.0% AN2690 Solution in the treatment of distal, subungual onychomycosis of the great target toenail.

DETAILED DESCRIPTION:
In this cohort, only the targeted great toenail identified at Baseline prior to the commencement of treatment from culture results collected at the Screening visit were evaluated for primary efficacy whereas all treated toenails were evaluated for safety. At each visit, the investigator was asked to make a clinical evaluation of the targeted great nail, marking whether or not they considered the nail to be clear of onychomycosis. This evaluation was the basis for determining whether or not study medication should be dispensed at the visit.

This record includes information only for Cohort 3 (5% solution) of the study. Cohorts 1 and 2, are described in NCT00679523 (7.5% solution). No comparison was made between Cohorts 1&2 and Cohort 3.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must meet all of the following criteria to be included in the study:
2. Witnessed, signed informed consent approved by Ethics Committee.
3. Male or female subjects of any race at least 18 years of age but not older than 65 years of age at the time of screening.
4. For Cohorts 1 and 2, subjects with a diagnosis of onychomycosis of at least one great toenail and with a positive KOH wet mount from that nail. For Cohort 3, subjects must have a diagnosis of onychomycosis of at least one great toenail and a positive KOH wet mount AND fungal culture from that nail.
5. Onychomycosis involving 20-60% of the affected great toenail as determined by visual inspection after the nail has been trimmed.
6. The combined thickness of the distal nail plate and the associated hyperkeratotic nail bed <3 mm.
7. Affected great toenail to be treated is capable of re-growth as documented by history or recent observation of at least 2 mm of growth.
8. Normal or not clinically significant screening safety labs.

Exclusion Criteria:

1. Females of childbearing potential not using a highly effective method of birth control (e.g. implants, injectables, combined oral contraceptives, some intrauterine contraceptive devices) during the study.
2. Diabetes mellitus requiring treatment other than diet and exercise.
3. Subjects with chronic moccasin type of T. pedis.
4. Subjects with a history of having failed any previous topical antifungal therapy for their onychomycosis.
5. Subjects unwilling to refrain from the use of nail cosmetics such as clear and or colored nail lacquers from the screening visit until the end of the study.
6. Subjects that have not undergone the specified washout period(s) for the following topical preparations or subjects who require the concurrent use of any of the following topical medications:

   * Topical antifungal applied to the feet (does not include antifungals for treatment of T. pedis during the study): 4 weeks
   * Anti-inflammatories, corticosteroids, topical immunomodulators: 2 weeks
7. Subjects that have not undergone the specified washout period(s) for the following systemic medications or subjects who require the concurrent use of any of the following systemic medications:

   * Corticosteroids (including intramuscular injections): 2 weeks
   * Antifungals for treatment of onychomycosis or any systemic antifungal with known activity against dermatophytes: 24 weeks
   * Systemic immunomodulators: 4 weeks
8. Treatment of any type for cancer within the last 6 months.
9. History of any significant internal disease.
10. Subjects with a medical history of current or past psoriasis of the skin and/or nails.
11. Concurrent lichen planus.
12. Subjects who are known to be allergic to any of the test product(s) or any components in the test product(s) or history of hypersensitivity or allergic reactions to any of the study preparations as described in the Investigator's Brochure.
13. Nail or anatomic abnormalities of the toe, e.g., genetic nail disorders, primentary disorders, onychogryphosis, trauma to the nail(s) to be treated.
14. AIDS or AIDS related complex.
15. History of street drug or alcohol abuse.
16. Any subject not able to meet the study attendance requirements.
17. Subjects who have participated in any other trial of an investigational drug or device within 60 days prior to enrollment or participation in a research study concurrent with this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Mexico (2):
  - Instituto Dermatologico Jalisciense, Guadalajara
  - IMIC, Mexico City

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled and two investigative sites in Mexico. The study population included men and women of any race, 18-65 years of age who had distal, subungual onychomycosis of the great toenail. The first subject visit occurred on March 28, 2007, and the last subject visit occurred on July 11, 2008.
Pre-assignment Details: All subjects in Cohort 3 were treated with 5.0% AN2690 Solution.
Period: Overall Study
Arm/Group | AN2690 Solution, 5.0%
Started | 29
Completed | 28
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: All analyses were performed using the intent-to-treat (ITT) population.
Arm/Group | AN2690 Solution, 5.0%
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 29
Age [Mean (Standard Deviation); unit: years] | 46.9 (10.15)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Evidence of Complete Clearance of the Treatment-targeted Great Toenail Plus a Negative Fungal Culture at Day 360
Description: Proportion of subjects with a clinical assessment of a clear (completely normal) nail unit plus a negative fungal culture from the treatment-targeted toenail at Day 360.
Time Frame: Day 360
Population: Efficacy data were analyzed for the ITT population. For efficacy variables, the last observation was carried forward (LOCF) to impute missing observations.
Measure: Number; unit: participants
Arm/Group | AN2690 Solution, 5.0%
Number analyzed (Participants) | 29
participants
  Success | 2 [0.0 to 16.1]
  Failure | 27

2. Secondary Outcome: Clear Nail Growth of the Targeted Toenail
Description: Clear nail was measured on digital images as the distance in millimeters from the proximal nail fold to the proximal limit of the disease as marked by the Investigator. New Clear Nail Growth (CNG) was calculated from the clear nail measurements.
Time Frame: Day 360
Population: Efficacy data were analyzed for the ITT population. For efficacy variables, the LOCF was used to impute missing observations.
Measure: Mean (95% Confidence Interval); unit: millimeters
Arm/Group | AN2690 Solution, 5.0%
Number analyzed (Participants) | 29
millimeters | 0.5 [-0.8 to 1.9]

3. Secondary Outcome: Mycological Evaluations (Negative Potassium Hydroxide (KOH) and Negative Fungal Culture) Compared to Baseline
Description: Number of subjects with negative KOH, and number of subjects with negative fungal cultures.
Time Frame: Day 90
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | AN2690 Solution, 5.0%
Number analyzed (Participants) | 29
participants
  Fungal Culture Result Positive | 1
  Fungal Culture Result Negative | 28 [89.9 to 100]
  KOH Result Positive | 24
  KOH Result Negative | 5 [3.5 to 31.0]

4. Secondary Outcome: Mycological Evaluations (Negative KOH and Negative Fungal Culture) Compared to Baseline
Description: Number of subjects with negative KOH, and number of subjects with negative fungal cultures.
Time Frame: Day 180
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | AN2690 Solution, 5.0%
Number analyzed (Participants) | 29
participants
  Fungal Culture Result Positive | 0
  Fungal Culture Result Negative | 29 [100 to 100]
  KOH Result Positive | 20
  KOH Result Negative | 9 [14.2 to 47.9]

5. Secondary Outcome: Mycological Evaluations (Negative KOH and Negative Fungal Culture) Compared to Baseline
Description: Number of subjects with negative KOH, and number of subjects with negative fungal cultures.
Time Frame: Day 270
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | AN2690 Solution, 5.0%
Number analyzed (Participants) | 29
participants
  Fungal Culture Result Positive | 1
  Fungal Culture Result Negative | 28 [89.9 to 100]
  KOH Result Positive | 17
  KOH Result Negative | 12 [23.5 to 59.3]

6. Secondary Outcome: Mycological Evaluations (Negative KOH and Negative Fungal Culture) Compared to Baseline
Description: Number of subjects with negative KOH, and number of subjects with negative fungal cultures.
Time Frame: Day 360
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | AN2690 Solution, 5.0%
Number analyzed (Participants) | 29
participants
  Fungal Culture Result Positive | 1
  Fungal Culture Result Negative | 28 [89.9 to 100]
  KOH Result Positive | 23
  KOH Result Negative | 6 [5.9 to 35.4]

7. Secondary Outcome: Length of Time to Clinical Evaluation of Clear or at Least 5 mm of CNG
Description: Length of time to clinical evaluation of clear or at least 5 mm of CNG.
Time Frame: Baseline to 360
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | AN2690 Solution, 5.0%
Number analyzed (Participants) | 29
days | 138.0 [81.5 to 194]

ADVERSE EVENTS:
Time Frame: Pre and post treatment to Day 360
Description: AEs were defined as any change (expected or unexpected) in a subject's medical health that occurred during the study. A serious AE was fatal, life-threatening, resulted in persistent or significant disability or incapacity, required or prolonged inpatient hospitalization, was a congenital anomaly, or another medically important condition.
Arm/Group | AN2690 Solution, 5.0%
Serious Adverse Events (participants affected / at risk) | 1/29
Other Adverse Events (participants affected / at risk) | 16/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AN2690 Solution, 5.0% (N=29)
Uterine haemorrhage (unrelated) (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AN2690 Solution, 5.0% (N=29)
Leukopenia (Blood and lymphatic system disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Abscess (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 7
Pyelonephritis (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Blood glucose abnormal (Investigations) | 1
Epilepsy (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Polycystic ovaries (Reproductive system and breast disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 1
Tooth extraction (Surgical and medical procedures) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution or Principal Investigator may only publish Study results after: (i) the results of the multicenter Study in its entirety have been publicly disclosed by the Sponsor in an abstract, manuscript or presentation form, or (ii) two (2) years after conclusion of the Study at all sites, whichever is first to occur.